CLINICAL TRIAL: NCT04757337
Title: Randomized Phase III Study of Oral Cyclophosphamide vs Doxorubicin in 65 Years or Older Patients With Advanced or Metastatic Soft Tissue Sarcoma: a UNICANCER/GERICO Multicenter Program
Brief Title: Comparison of Oral Cyclophosphamide vs Doxorubicin in ≥65 Years Old Advanced or Metastatic Soft Tissue Sarcoma Patients
Acronym: GERICO14
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0103/1802; 2018-000542-20 (EudraCT Number)
Record Dates: First submitted 2021-02-10; First posted 2021-02-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-06

CONDITIONS: Advanced Soft-tissue Sarcoma; Metastatic Soft-tissue Sarcoma
Keywords: Elderly; older patients; oral cyclophosphamide; doxorubicin
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxorubicin (Active Comparator): Intravenous Doxorubicin 60 mg/m² Cycle 1 then 75 mg/m² Cycle 2 to Cycle 6 D1-D21 with granulocyte-colony stimulating factor (G-CSF) and dexrazoxane.
  Interventions: Drug: Doxorubicin
- Cyclophosphamide (Experimental): Cyclophosphamide per os 100 mg twice a day, 1 week on, 1 week off until 2 years, or unacceptable toxicity, disease progression, withdrawn of consent or death.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Doxorubicin — 6 x 3-week cycles corresponding to a maximal duration of 18 weeks
  Arms: Doxorubicin
Drug: Cyclophosphamide — Until progression up to 24 months
  Other Names: Endoxan®
  Arms: Cyclophosphamide

SUMMARY:
Most advanced or metastatic soft tissue sarcoma (STS) are unfortunately incurable, making the preservation of the patient's quality of life a major goal, along with prolonging survival.

Age is not a criterion for not providing effective treatment, but the goals of treatment change with age and must be integrated into the treatment decision. Elderly patients prioritise a life free of dependency, preservation of their cognitive functions and quality of life related to their state of health. They are therefore reluctant to receive a treatment that does little to improve life expectancy at the cost of significant functional losses.

Patients aged 65 years and older account for one third of all patients with STS. In the absence of dedicated recommendations, these elderly patients are currently receiving doxorubicin-based chemotherapy as first-line treatment (as recommended for younger patients), with a substantial risk of toxicity (especially cardiac). In this specific population, previous studies have shown that oral cyclophosphamide seems to have a promising activity, but also a very acceptable toxicity.

Thus, the GERICO study aims to compare standard doxorubicin chemotherapy with oral cyclophosphamide for the treatment of elderly patients with STS.

DETAILED DESCRIPTION:
Co-morbidities increase in number and severity with age, competing with cancer prognosis and making prioritizing medical issues necessary. Individualization of cancer treatment by integrating a comprehensive geriatric assessment (CGA) is frequently considered as essential and mandatory for elderly cancer patients. The G8 questionnaire is able to identify patients requiring CGA, with a threshold score of ≤14/17 and with a strong 1-year prognostic value.

According to guidelines, the recommended first-line treatment of these patients relies on single agent chemotherapy with anthracyclines (including doxorubicin); however, anthracycline-based treatments have modest performance in patients with metastatic STS with a median progression-free survival of about 4 months and an overall survival of about 12 months.

Previous studies have demonstrated promising activity of oral metronomic cyclophosphamide in STS patients and its favorable safety profile.

To evaluate this promising activity we designed a phase III, randomized, open-label, multicentric study comparing daily oral cyclophosphamide versus standard 3-week intravenous injection of doxorubicin in 65 years or older patients with advanced or metastatic STS.

ELIGIBILITY:
Inclusion criteria:

1. Patient must have signed a written informed consent form prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trust person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent
2. Age ≥65 years (inclusions will be managed to ensure that at least 50% of the randomized patients are ≥75 years old)
3. Diagnosis of soft-tissue sarcoma histologically confirmed by Réseau de Référence en Pathologie des Sarcomes et des Viscères (RRePS)
4. Metastatic or locally advanced disease not amenable to surgery, radiation, or combined modality treatment with curative intent. Palliative radiation therapy is permitted only if direct on nontarget lesion
5. Documentation of disease progression within the last 6 months before randomization
6. Measurable disease, defined as at least 1 unidimensionally measurable lesion on a CT-scan as defined by response evaluation criteria in solid tumors version 1.1 (RECIST v1.1)
7. Life expectancy of at least 6 months
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤2
9. G8 score >14
10. Left ventricular ejection fraction (LVEF) value by echocardiogram or Multiple gated acquisition scanning (MUGA) ≥55%
11. Adequate bone marrow, renal, and hepatic function, as evidenced by the following within 7 days of study treatment initiation:

    1. Absolute neutrophil count (ANC) ≥1,500/mm³
    2. Platelets ≥100,000/mm³
    3. Hemoglobin ≥9.0 g/dL
    4. Serum creatinine ≤2 x upper limit of normal (ULN)
    5. Glomerular filtration rate (GFR) ≥50 ml/min/1.73m² (calculated with MDRD)
    6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN (≤5.0 × ULN for patients with liver involvement of their cancer )
    7. Total bilirubin ≤1.5 X ULN
    8. Alkaline phosphatase ≤2.5 x ULN (≤5 x ULN with liver involvement of their cancer)
    9. serum albumin >25 g/L
    10. Prothrombin time (PT)/International normalized ratio (INR) ≤1.5 x ULN Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until PT/INR is stable based on a measurement that is pre-dose as defined by the local standard of care
12. Male patients must agree to use adequate contraception for the duration of trial participation and up to 6 months after completing treatment/therapy. Adequate contraception is defined as any medically recommended method (or combination of methods) as per standard of care
13. Patients must be affiliated to a Social Security System (or equivalent)
14. Patient is willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures including follow-up

Exclusion Criteria:

1. Previous systemic treatment for advance or metastatic sarcoma
2. Previous neoadjuvant or adjuvant anthracycline treatment for localized sarcoma
3. Soft-tissue sarcoma with the following histological subtypes: dermatofibrosarcoma protuberans, desmoid tumor, alveolar or embryonal rhabdomyosarcoma, Desmoplastic small round cell tumor, Kaposi Sarcoma, Gastro-Intestinal stromal tumor, Peripheral neuroectodermal tumors
4. Primary bone sarcoma (including osteosarcoma, Ewing tumor, chondrosarcoma, and chordoma)
5. Symptomatic or known central nervous system (CNS) metastases
6. Known history of or concomitant malignancy likely to affect life expectancy in the judgment of the investigator and history of radiotherapy mediastinal in the last five years
7. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before Day 1 of treatment
8. Active cardio vascular disease including any of the following: Congestive heart failure (New York Heart Association (NYHA) ≥Class 2), unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months), acute inflammatory cardiopathy, severe arrythmia, high risk of bleeding, cerebrovascular accident within the last 6 months
9. Uncontrolled grade >2 hypertension. (Systolic blood pressure ≥160 mmHg or diastolic pressure ≥100 mmHg despite optimal medical management)
10. Ongoing infection ≥Grade 2 according to NCI Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)
11. Known history of human immunodeficiency virus (HIV) infection
12. Known history of chronic hepatitis B or C
13. History of organ allograft
14. Pre-existing acute hemorrhagic cystitis, urinary tract obstruction, acute urinary tract infection
15. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
16. Substance abuse, medical condition, that may interfere with the patient's participation in the study or evaluation of the study results
17. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
18. Inability to swallow oral medications, any malabsorption condition.
19. Persons deprived of their liberty or under protective custody or guardianship
20. Participation in another therapeutic trial within the 30 days prior to randomization and during the study
21. Patients having received live attenuated vaccine therapy used for prevention of diseases as influenza, chickenpox, zoster, measles, mumps, rubella, tuberculosis, rotavirus or yellow fever within 4 weeks of the first dose of study drug. These vaccinations are not permitted during the study up to 6 months after the last treatment
22. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to disease progression or death, up to 2 years.
  The progression-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, up to 2 years
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Best response under treatment | From randomization to progression, death or new treatment, up to 2 years.
  Best response under treatment: Best response (as per RECIST v1.1) recorded from the date of randomization until the end of treatment. Each patient will be assigned one of the following categories: complete response, partial response, stable disease, disease progression, or unevaluable for response (specify reasons, e.g. early death, malignant disease; toxicity; tumor assessment not repeated/incomplete; other). Responses will have to be confirmed at least 4 weeks after the evaluation to exclude measurement errors.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, week 9, week 18, 3 months, 6 months, 9 months, 12 months, 15 month, 18 month, and 24 months
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire - Elderly cancer patients (QLQ-ELD14) | At baseline, week 9, week 18, 3 months, 6 months, 9 months, 12 months, 15 month, 18 month, and 24 months
  The EORTC QLQ-ELD14, a validated HRQOL questionnaire for cancer patients aged greater than or equal to70 years, is intended to supplement the QLQ-C30.
  The QLQ-ELD14 contains 14 items incorporating five scales to assess mobility, worries about others, future worries, maintaining purpose, and illness burden. In addition, two single items assess joint stiffness and family support. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. High scores indicate poor mobility, good family support, much worry about the future, good maintenance of autonomy and purpose, and high burden of illness.
Assessment of the toxicity profile of oral cyclophosphamide and doxorubicin, as per NCI CTCAE v5.0 | From randomization to progression, death or new treatment, up to 2 years.
  Toxicity: Adverse events will be graded according to the CTCAE v5.0.
Geriatric assessment | At baseline
  The Geriatric Core Dataset (G-CODE) was developed by the DIalog for personALization of management in geriatric OncoloGy (DIALOG) intergroup to assess the general health status of the older patient.
  The G-Code contains 10 tools incorporating seven scales to assess social environment, functional status, mobility, nutritional status, cognitive status, depressive mood, and comorbidities. The total scale range 0-62. High score indicate better condition.
Assessment of compliance to oral metronomic cyclophosphamide (Cyclophosphamide Arm only) | From randomization to the end of treatment, up to 2 years.
  Compliance to oral metronomic cyclophosphamide will be assessed based on data reported by the patients (patient diary).

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud Valentin, M.D, Principal Investigator — Institut Claudius Regaud-IUCT Oncopôle Toulouse; Olivier Mir, M.D, Principal Investigator — Gustave Roussy Cancer Institute
Locations (1):
- Institut Claudius Reagaud-IUCT Oncopôle, Toulouse, France

IPD SHARING:
Plan to Share IPD: No